CLINICAL TRIAL: NCT04826393
Title: Phase Ib Trial of ASP8374 and Cemiplimab in Recurrent Malignant Glioma Patients
Brief Title: ASP8374 + Cemiplimab in Recurrent Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, David Reardon, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-054
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma; Recurrent Glioblastoma
Keywords: Glioblastoma; Recurrent Glioblastoma; Glioma, Grade 3
MeSH Terms: conditions — Glioblastoma; Glioma; Lymphoma, Follicular | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ASP8374 and Cemiplimab-Cohort 1 (Experimental): A 3+3 dose escalation design will be used to determine maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of ASP8374 when combined with cemiplimab.
  Participants will receive ASP8374 and Cemiplimab every 3 weeks for up to 2 years. ASP8374 will be available until October 31, 2022. Subjects may continue treatment with cemiplimab alone after that date.
  Interventions: Drug: ASP8374; Drug: cemiplimab
- ASP8374 and Cemiplimab-Cohort 2 (Experimental): Upon determination of the MTD/RP2D of ASP8374 plus cemiplimab in Cohort 1, a dose expansion will be performed in which eligible participants who are candidates for surgical resection will enroll to Cohort 2 and will be randomized into one of two treatment groups (2A-2B).
  Group 2A: IV ASP8374 plus cemiplimab within 14± 5 days prior to surgery at the MTD/RP2D established in Cohort 1.
  Group 2B: No immune checkpoint therapy prior to surgery.
  Post-operatively, all Cohort 2 participants will receive ASP8374 plus cemiplimab every 3 weeks administered at the MTD/RP2D established by Cohort 1
  Interventions: Drug: ASP8374; Drug: cemiplimab

INTERVENTIONS:
Drug: ASP8374 — every 3 weeks by intravenous infusion
Drug: cemiplimab — intravenous infusion
  Other Names: Libtayo

SUMMARY:
This study is looking at the safety and efficacy of the drug combination of ASP8374 with cemiplimab in people with recurrent malignant glioma.

The study will be conducted in two parts, the first portion of the study will be to establish the highest dose of ASP8374 that can be given safely with cemiplimab and will be used as the recommended dose of ASP8374 in combination with cemiplimab for the second portion of the study. The second portion of the study will be to compare the effect of having ASP8374 in combination with cemiplimab prior to surgery.

The names of the study drugs involved in this study are:

* ASP8374
* Cemiplimab

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, phase Ib trial of ASP8374 plus cemiplimab among recurrent malignant glioma participants.

Initially, eligible participants will enroll to Cohort 1 which will determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of ASP8374 when combined with cemiplimab among recurrent malignant glioma participants using a 3+3 design.

Upon determination of the MTD/RP2D of ASP8374 plus cemiplimab in Cohort 1, a dose expansion will be performed in which eligible participants who are candidates for surgical resection will enroll to Cohort 2 and will be randomized into one of two treatment groups (2A-2B).

Group 2A: IV ASP8374 plus cemiplimab within 14± 5 days prior to surgery at the MTD/RP2D established in Cohort 1.

Group 2B: No immune checkpoint therapy prior to surgery.

The U.S. Food and Drug Administration (FDA) has not approved ASP8374 as a treatment for any disease. The U.S. Food and Drug Administration (FDA) has not approved cemiplimab for recurrent malignant glioma but it has been approved for other uses.

The research study procedures include: screening for eligibility, then study treatment including evaluations and follow up visits. Participants will receive study treatment for up to two years and will be followed for their tumor's response, whether or not their disease gets worse, and for side effects.

It is expected that about 24 people will take part in this research study. At least 6 in cohort 1 and 18 in cohort 2.

Pharmaceutical company Astellas is supporting this research study by providing study funding and study drug, ASP8374 and Regeneron is supporting this research by providing study drug cemiplimab.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed WHO grade IV GBM or its variants. Participants will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of GBM is made. Participants with WHO grade III recurrent malignant glioma will be allowed to enroll to Cohort 1 only.
* Be willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Have a Karnofsky performance status (KPS) ≥ 70 (Appendix A).
* Previous first line therapy with at least radiotherapy.
* Be at first or second relapse. Note: Relapse is defined as progression following initial therapy (i.e., radiation ± chemotherapy). For participants who had prior therapy for a low-grade glioma, the surgical diagnosis of a high-grade glioma will be considered the first relapse.
* Participants must have shown unequivocal evidence for tumor progression by MRI or CT scan.
* Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 14 days of registration.

  * Table 1: Adequate Organ Function Laboratory Values

    * System Laboratory Value

      * Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
      * Renal Serum creatinine OR measured or calculated a creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X institutional upper limit of normal (ULN) OR

        ≥60 mL/min for participant with creatinine levels > 1.5 X institutional ULN a Creatinine clearance should be calculated per institutional standard.
      * Hepatic Serum total bilirubin ≤ 1.5 X institutional ULN OR Direct bilirubin ≤ institutional ULN for participants with total bilirubin levels > 1.5 institutional ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X institutional ULN OR

        ≤ 5 X institutional ULN for participants with Gilberts syndrome Albumin >2.5 mg/dL
      * Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5 X institutional ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 X institutional ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Contrast enhanced CT or MRI within 14 days prior to registration. NOTE: For Cohort 2 participants only: due to the fact that the screening MRI will not be used for response purposes, participants may be registered if the screening scan is >14 days from registration with prospective approval from Overall PI, Dr. David Reardon (for prospectively approved circumstances, an eligibility exception will not need to be filed).
* An interval of at least 3 weeks (to registration) between prior surgical resection or one week for stereotactic biopsy.
* An interval of at least 12 weeks from the completion of radiation therapy to registration unless there is unequivocal histologic confirmation of tumor progression or radiographic progression outside of the prior radiation field.
* Participants must have recovered to grade 0 or 1 or pre-treatment baseline from clinically significant toxic effects of prior therapy (exceptions include but not limited to alopecia, laboratory values not listed per inclusion criteria, and lymphopenia which is common after therapy with temozolomide).
* From start of study therapy, the following time periods must have elapsed:

  * 5 half-lives from any small molecule investigational agent
  * 4 weeks from cytotoxic therapy (except 23 days for temozolomide, 6 weeks from nitrosoureas, and 7 days from daily administered agents)
  * 6 weeks from antibodies, or 4 weeks (or 5 half-lives, whichever is shorter) from other anti-tumor therapies
  * No wash-out period required for prior TTF or vaccine therapies
* Participants must be planned to undergo surgery that is clinically indicated as determined by their care providers (Cohort 2 only).
* Female participant of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment she considered not of child bearing potential.
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during study treatment and for 120 days after study discontinuation. Highly effective contraception is defined as either:

  * i. True Abstinence: When this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * ii. Sterilization: Surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment (as described in item 12 above).
  * iii. Male Partner Sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female participants on the study, the vasectomized male partner should be the sole partner for that participant.
  * Use of a combination of any two of the following:

    1. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    2. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
    3. Appropriate hormonal contraceptives (including any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent - including oral, subcutaneous, intrauterine, or intramuscular agents)
* Male participants should agree to use adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of therapy.

Exclusion Criteria:

* Current or planned participation in a study of an investigational agent or using an investigational device.
* Has a diagnosis of immunodeficiency.
* Has tumor primarily localized to the brainstem or spinal cord.
* Has presence of diffuse leptomeningeal disease or extracranial disease.
* Has received systemic immunosuppressive treatments, aside from systemic corticosteroids as described in Section 3.2.7, (such as methotrexate, chloroquine, azathioprine, etc.) within six months of registration.
* Has received anti-VEGF or anti-VEGFR targeted agents (e.g. bevacizumab, cediranib, aflibercept, vandetanib, XL-184, sunitinib, etc.).
* Requires treatment with moderate or high dose systemic corticosteroids defined as dexamethasone > 2 mg/day or bioequivalent for at least 3 consecutive days within 7 days of registration.
* Has received prior interstitial brachytherapy or stereotactic radiosurgery (Cohort 2 only).
* Has history of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 12 months of registration.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE Grade > 3 within 6 months of registration.
* Has a known additional malignancy that is progressing or requires active treatment within 2 years of registration. Exceptions include malignancies treated with surgery alone including but not limited to basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. See Section 5.4.3 for additional information on allowed corticosteroid dosing.
* Has confirmed history or any evidence of active non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator. Examples include but are not limited to symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment. It is unknown whether ASP8374 and/or cemiplimab is excreted in human milk or may have adverse effects on a fetus in utero. Since many drugs are excreted in human milk, and because of the potential for serious adverse reactions in the nursing infant or fetus, these participants are not eligible for enrollment.
* Has received prior therapy with an anti-TIGIT, anti-PD-1, anti-PD-L1, anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab), or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days prior to registration.
* Has a known hypersensitivity to any of the study therapy products.
* Has been previously treated with the PI3K inhibitor idelalisib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Maxium Tolerated Dose-MTD/ Phase 2 Recommend Dose-RP2D - Cohort 1 | Enrollment up to 2 years
  primary endpoint for Cohort 1 will be determination of the MTD/RP2D of ASP8374 when administered with cemiplimab among recurrent malignant glioma participants.
CD8+ TIL Tumor Density-Cohort 2 | Enrollment up to 2 years
  CD8+ TIL density from tumors obtained from participants randomized to the neoadjuvant study arm (2A) will be compared to tumor CD8+ TIL density obtained from control participants enrolled on Arm 2B who do not receive neoadjuvant therapy.

SECONDARY OUTCOMES:
Rate of Adverse Events | Enrollment up to 2 years
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
progression-free survival (PFS) | 6 months
  Assessed by Response Assessment in Neuro-Oncology (RANO)1 and Immunotherapy RANO (iRANO) guidelines.
overall survival (OS). | 12 months
  Assessed by Response Assessment in Neuro-Oncology (RANO)1 and Immunotherapy RANO (iRANO) guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: David A Reardon, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Hospital of the University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu